CLINICAL TRIAL: NCT04179734
Title: Physiological Study to Determine the Role of the Melanocortin-4 Receptor in Brain Activity in Women With Hypoactive Sexual Desire Disorder
Brief Title: Role of the Melanocortin-4 Receptor in Hypoactive Sexual Desire Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 262886
Record Dates: First submitted 2019-11-01; First posted 2019-11-27 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: Hypoactive Sexual Desire Disorder; Bremelanotide; Functional MRI; Melanocortin-4 receptor
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — bremelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Bremelanotide 1.75 mg - prefilled subcutaneous autoinjector containing 1.75 mg Bremelanotide in a 0.3 mL solution volume.
  Interventions: Drug: Bremelanotide; Drug: Placebo
- Placebo (Placebo Comparator): 1.75 mg equivalent - prefilled subcutaneous autoinjector containing Bremelanotide formulation without the active ingredient in a 0.3 mL solution volume.
  Interventions: Drug: Bremelanotide; Drug: Placebo

INTERVENTIONS:
Drug: Bremelanotide — Melanocortin-4 receptor agonist subcutaneous injection.
Drug: Placebo — Placebo subcutaenous injection.

SUMMARY:
A randomised, double-blind, placebo-controlled, two-way crossover physiological study. Designed to evaluate the effects of melanocortin-4 receptor (MC4R) activation on brain activity patterns and behavioural psychometric measures of sexual arousal during visual erotic stimuli in approximately 40 right-handed, heterosexual, premenopausal women aged 18 years and over with Hypoactive Sexual Desire Disorder (HSDD) for at least a 6 month duration.

DETAILED DESCRIPTION:
The investigators aim to recruit approximately 40 women to allow for subject and technical drop-out, aiming for a minimum of 30 women in the final study who complete the full protocol successfully. The investigators will collaborate with the Sexual Medicine clinic to identify potential participants, as well as advertise via print (including local and regional newspapers, transport network), radio and online advertisements. Additionally, the investigators will liaise with the local Clinical Research Network (CRN) to contact potentially eligible patients via their General Practitioner (GP) surgery (via letter or text message). Potential participants who contact us via advertisements will initially be electronically sent a participant information sheet and self-report questionnaire, to be returned via email. If, following this, they are happy to take part and no obvious exclusion criteria are detected, they will be screened via telephone using a questionnaire. If eligible, they will be invited for a formal screening interview, where further questions regarding the study will be answered. After obtaining consent, a full medical and sexual history will be taken as well as a review of the diagnosis of assessment, an ECG, urinalysis to exclude pregnancy, clinical laboratory testing and completion of psychiatric and psychosexual questionnaires.

Eligible participants will then enter the Intervention phase. Participants will be randomised (1:1) to one of two intervention sequences: a single dose of Bremelanotide or matching placebo, administered subcutaneously. All participants will attend for two study visits each, during which they will undergo a functional magnetic resonance imaging (fMRI) scan while receiving either Bremelanotide or placebo. During the scan, participants will be presented with visual erotic stimuli in order to activate the brain, so that Bremelanotide's modulation of the melanocortin system can be measured. The participants will also be asked to use a behavioural potentiometer whilst in the scanner to rate their degree of sexual arousal. The crossover design, which allows participants to serve as their own control, will minimise inter-participant variability. Participants will also be sent a short questionnaire 24-hours after the study to assess the perceived duration of effect of Bremelanotide.

The MRI data will be processed and analysed using current best practice methods, which will include (but may not be limited to) application of the General Linear Model (GLM) for neuroimaging data. Robust methods of correcting for multiple comparisons (e.g. permutation testing) will be used for statistical analysis and thresholding of the statistical brain images. Brain activation patterns will be presented by intervention and analysed by whole-brain and region of interest (including amygdala, thalamus, posterior cingulate cortex and entorhinal region. Correlations will be explored between brain activation and behavioural data, corrected for visit order as appropriate (including Pearson and Partial Correlation testing).

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual premenopausal females ≥ 18 years of age with normal menstrual cycles ≤ 35 days.
* Right hand dominant.
* Body mass index (BMI) 18-35kg/m2.
* Currently in a relationship with a male partner and the relationship has been stable for at least 6 months before screening.
* Male sexual partner classified as "not impotent" on the Massachusetts Male Aging Study (MMAS) single-question assessment of erectile dysfunction.
* In the subject's opinion, previously experienced "normal sexual function," defined as a normal level of desire at some point in the past, for a period of at least 2 years.
* For all subjects of childbearing potential who are sexually active, agree to routinely use adequate non-hormonal contraception from randomisation throughout the duration of the study and for 30 days after.
* For at least 6 months before Screening, met the diagnostic criteria for HSDD according to the Diagnostic Screening Guide for HSDD, including categorisation of the sexual dysfunction as both acquired (versus lifelong) and generalised (versus situational).
* All of the following at Screening:

  1. Patient Health Questionnaire (PHQ-9) (Kroenke et al., 2001) total score is <10.
  2. PHQ-9 score for Question 9 is 0.

  <!-- -->

  1. Either Female Sexual Function Index (FSFI) total score ≤26 if diagnosed with HSDD (with or without symptoms of decreased arousal) or subjects diagnosed with HSDD only (without symptoms of decreased arousal), FSFI desire domain score of ≤5 (regardless of total FSFI score).
  2. Female Sexual Distress Scale - Desire/Arousal/Orgasm (FSDS-DAO) total score is >18.
* Capable of understanding and complying with the protocol requirements and available for the duration of the study.
* Subjects must have prior experience in viewing sexually explicit material.

Exclusion Criteria:

* Cardiovascular disease
* Current diagnosis of uncontrolled hypertension defined as:

  1. Two sequential assessments (seated, approximately 4 minutes apart and no more than 15 minutes apart) with readings above 140 mmHg systolic BP or 90 mmHg diastolic BP, and upon repeat at least 24 hours later.
  2. Treatment for hypertension that has been changed at least once in the 4 weeks prior to Screening.
* Any other medical condition that is unstable or uncontrolled despite current therapy.
* Previously received Bremelanotide.
* A history of unresolved sexual trauma or abuse.
* Female subjects who are pregnant, intend to become pregnant, are breastfeeding, have a positive serum/urine pregnancy test, or are not willing to use effective contraceptive precautions during the study.
* Participated in any research study within the preceding 30 days of screening.
* Any FSD other than acquired HSDD with or without decreased arousal (e.g. lifelong anorgasmia, sexual pain disorder, sexual aversion disorder, primary female sexual arousal disorder).
* FSD caused by untreated endocrine disease (e.g. hypopituitarism, hypothyroidism, diabetes mellitus).
* Acute or chronic hepatitis.
* In the Investigator's opinion, any urologic or gynecologic condition, such as condyloma, uterine fibroids, vulvar or vaginal lesions, vulvodynia, vaginismus, or pelvic pain that may contribute to impaired sexual activity and function or be a cause of the FSD or that may interfere with the subject's ability to comply with study procedures.
* Receiving any treatment for HSDD (e.g. psychotherapy, physical therapy) at the time of Screening.
* Has used any of the following types of medications, which are prohibited during the study:

  1. Implanted or injected testosterone product within 6 months of Screening.
  2. Within 3 months of Screening:
* Neuroleptics (e.g. risperidone)
* Lithium (e.g. lithium carbonate)
* Antidepressants (e.g. amitriptyline, fluoxetine, bupropion)
* Mood stabilisers (e.g. valproate)
* Benzodiazepines (e.g. lorazepam, diazepam)
* Cognitive enhancers or stimulants (e.g. donepezil or Adderall®)
* Centrally-acting antihypertensives (e.g. clonidine)
* Any other prescription, non-prescription, hormonal, herbal, or nutritional medication or supplement that the investigators believe would confound the results of the study (e.g. St. John's wort, black cohosh, dehydroepiandrosterone, dehydroepiandrosterone sulfate)
* γ-Aminobutyric acid agonists (e.g. Ambien® [zolpidem], Lunesta® [eszopiclone]) c. Topical or systemic androgen therapy within 30 days of Screening. d. Subject is unwilling or unable to refrain from using the aforementioned products for the duration of the study.
* Mental health history that includes any of the following:

  1. Psychosis, bipolar disorder, depression, and/or alcohol/substance abuse; depression or alcohol/substance abuse that resolved >1 year prior to Screening/Visit 1 will not be exclusionary.
  2. Prior suicide attempt or increased suicidality as indicated by a score greater than zero on Questions 1-5 inclusive (interpreted increased risk) and/or Question 20 (interpreted history of suicide) of the Beck Scale for Suicidal Ideation (BSS),
* Any abnormality in vision that would impair viewing images.
* Any contraindication to MRI or otherwise unable to undergo an MRI (e.g. pacemaker, recent wound clips, severe claustrophobia, unable to lay flat).
* Any other condition or subject responsibility that in the Investigator's opinion may interfere with a subject's ability to give informed consent or adhere to the protocol or has the potential to interfere with the studied endpoints or serves as a contraindication to the subject's participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waljit S Dhillo, MBBS PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnow BA, Millheiser L, Garrett A, Lake Polan M, Glover GH, Hill KR, Lightbody A, Watson C, Banner L, Smart T, Buchanan T, Desmond JE. Women with hypoactive sexual desire disorder compared to normal females: a functional magnetic resonance imaging study. Neuroscience. 2009 Jan 23;158(2):484-502. doi: 10.1016/j.neuroscience.2008.09.044. Epub 2008 Oct 2. PMID 18976696
- [Background] Bianchi-Demicheli F, Cojan Y, Waber L, Recordon N, Vuilleumier P, Ortigue S. Neural bases of hypoactive sexual desire disorder in women: an event-related FMRI study. J Sex Med. 2011 Sep;8(9):2546-59. doi: 10.1111/j.1743-6109.2011.02376.x. Epub 2011 Jun 30. PMID 21718449
- [Background] Pfaus JG, Shadiack A, Van Soest T, Tse M, Molinoff P. Selective facilitation of sexual solicitation in the female rat by a melanocortin receptor agonist. Proc Natl Acad Sci U S A. 2004 Jul 6;101(27):10201-4. doi: 10.1073/pnas.0400491101. Epub 2004 Jun 28. PMID 15226502
- [Background] Shifren JL, Monz BU, Russo PA, Segreti A, Johannes CB. Sexual problems and distress in United States women: prevalence and correlates. Obstet Gynecol. 2008 Nov;112(5):970-8. doi: 10.1097/AOG.0b013e3181898cdb. PMID 18978095
- [Background] Murphy K, Garavan H. An empirical investigation into the number of subjects required for an event-related fMRI study. Neuroimage. 2004 Jun;22(2):879-85. doi: 10.1016/j.neuroimage.2004.02.005. PMID 15193618
- [Background] Wikberg JE, Muceniece R, Mandrika I, Prusis P, Lindblom J, Post C, Skottner A. New aspects on the melanocortins and their receptors. Pharmacol Res. 2000 Nov;42(5):393-420. doi: 10.1006/phrs.2000.0725. PMID 11023702
- [Background] Woodard TL, Nowak NT, Balon R, Tancer M, Diamond MP. Brain activation patterns in women with acquired hypoactive sexual desire disorder and women with normal sexual function: a cross-sectional pilot study. Fertil Steril. 2013 Oct;100(4):1068-76. doi: 10.1016/j.fertnstert.2013.05.041. Epub 2013 Jul 2. PMID 23830149
- [Background] Kingsberg SA, Clayton AH, Portman D, Williams LA, Krop J, Jordan R, Lucas J, Simon JA. Bremelanotide for the Treatment of Hypoactive Sexual Desire Disorder: Two Randomized Phase 3 Trials. Obstet Gynecol. 2019 Nov;134(5):899-908. doi: 10.1097/AOG.0000000000003500. PMID 31599840
- [Result] Thurston L, Hunjan T, Mills EG, Wall MB, Ertl N, Phylactou M, Muzi B, Patel B, Alexander EC, Suladze S, Modi M, Eng PC, Bassett PA, Abbara A, Goldmeier D, Comninos AN, Dhillo WS. Melanocortin 4 receptor agonism enhances sexual brain processing in women with hypoactive sexual desire disorder. J Clin Invest. 2022 Oct 3;132(19):e152341. doi: 10.1172/JCI152341. PMID 36189794

RESULTS

PARTICIPANT FLOW:
Groups:
- Bremelanotide First, Then Placebo: Participants attended 2 study visits each: first visit (6 hours) for subcutaneous administration of Bremelanotide 1.75 mg/0.3 mL then at least one month later a second visit (6 hours) for subcutaneous administration of equivalent volume Placebo. This was to ensure full washout between visits and to allow the study to be performed at the same stage of the participant's menstrual cycle each time.
- Placebo First, Then Bremelanotide: Participants attended 2 study visits each: first visit (6 hours) for subcutaneous administration of equivalent volume Placebo then at least one month later a second visit (6 hours) for subcutaneous administration of Bremelanotide 1.75 mg/0.3 mL. This was to ensure full washout between visits and to allow the study to be performed at the same stage of the participant's menstrual cycle each time.
Period: Group 1 Bremelanotide, Group 2 Placebo
Arm/Group | Bremelanotide First, Then Placebo | Placebo First, Then Bremelanotide
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Group 1 Placebo, Group 2 Bremelanotide
Arm/Group | Bremelanotide First, Then Placebo | Placebo First, Then Bremelanotide
Started | 20 | 20
Completed | 16 | 15
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Abnormal structural findings on MRI | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bremelanotide First, Then Placebo | Placebo First, Then Bremelanotide | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [25 to 36] | 29 [25 to 36] | 29 [25 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Changes in Blood Oxygen Level Dependent (BOLD) Signal Change on Functional MRI
Description: Blood Oxygen Level Dependent (BOLD) imaging was used to detect activation clusters within the brain. Units of measure were standardised regression coefficients derived from the regression analysis that were used to fit the analysis model to the time-series data (BOLD signal change). Higher BOLD signal change values indicate increased activation in particular areas of the brain in response to the intervention (Bremelanotide or Placebo).
Time Frame: Baseline and 15 minutes
Population: A final group of 31 premenopausal women with HSDD participated in a randomized, double-blinded, 2-way crossover, placebo- controlled study. They attended 2 study visits each: 1 for subcutaneous administration of Bremelanotide and 1 for subcutaneous administration of an equivalent volume of placebo in random order, at least 1 month apart.
Measure: Number; unit: BOLD signal change
Groups:
- Bremelanotide: Participants were administered a subcutaneous injection of the melanocortin-4 receptor agonist (MC4Ra) Bremelanotide.
- Placebo: Participants were administered a subcutaneous injection of equivalent volume of placebo.
Arm/Group | Bremelanotide | Placebo
Number analyzed (Participants) | 31 | 31
BOLD signal change | 9.98 | 7.67

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the two 6-hour study visits which were at least one month apart (mean, 1.32; SEM, 0.12).
Groups:
- Bremelanotide: All 31 participants received Bremelanotide. 16 participants received Bremelanotide on their first study visit and 15 participants received Bremelanotide on their second study visit in this randomized, double-blinded, 2-way crossover study.
- Placebo: All 31 participants received Placebo. 15 participants received Placebo on their first study visit and 16 participants received Placebo on their second study visit in this randomized, double-blinded, 2-way crossover study.
Arm/Group | Bremelanotide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT04179734/Prot_SAP_000.pdf